CLINICAL TRIAL: NCT01997203
Title: Effect of Long-term Vitamin D Therapy on IL-6, Visfatin and Hyaluronic Acid in Hepatitis C Virus Patients' Assessment
Brief Title: Long Term Vitamin D Therapy in HCV Treated Patients
Acronym: VD-HCV
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: complete patients samples required
Sponsor: Dr. Nadia AbdelAaty AbdelKader (Other)
Responsible Party: Sponsor-Investigator, Dr. Nadia AbdelAaty AbdelKader, Ass. prof. Tropical Medicine - Ain Shams University, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCV-VD2013
Record Dates: First submitted 2013-11-19; First posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Hepatitis C
Keywords: hepatitis C infection; vitamin D
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Vitamin D; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HCV patients under treatment (Experimental): Fifty patients study group administered vitamin D were compared with 50 patients control group without vitamin D.
  Dose of vitamin D 15,000 IU/week
  Interventions: Drug: Vitamin D
- HCV without Vit D (No Intervention)

INTERVENTIONS:
Drug: Vitamin D — vitamin D was given to 50 patients (HCV under treatment)
  Other Names: pegylated interferon; ribavirin
  Arms: HCV patients under treatment

SUMMARY:
Treatment of hepatitis C virus (HCV) infection was carried out using pegylated interferon (PEG-IFN), ribavirin (RBV) and vitamin D (vit D) for 48 weeks in HCV genotypes 4a subjects. The purpose of this study is to determine the effect of vitamin D on liver affection in such patients.

DETAILED DESCRIPTION:
Fifty patients study group administered vit D were compared with 50 patients control group without vit D. The results showed a significant elevation in vit D levels during the time period, and significant reduction on HCV RNA from the 12th wk to reach zero level in 24th wk. Interleukin 6 (IL-6), visfatin and hyaluronic acid levels were reduced significantly to reach normal values. These concentrations reduction by the effect of vit D on HCV indicated the reduction in inflammation, infection and liver cirrhosis and nearly amelioration HCV.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV infection (positive HCV Ab more than 6 months)
* Treated with pegylated interferon and ribavirin

Exclusion Criteria:

* Coinfection with Hepatitis B or Hepatitis D or Human Immunodeficiency Virus
* Previous non response to antiviral therapy.
* Other causes of chronic liver diseases as schistosomiasis, Wilson disease and alcoholic liver disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
composite measures of Vitamin D, IL-6, Visfatin and Hyaluronic acid in Hepatitis C Virus Patients under antiviral therapy | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dina Sabry, Principal Investigator — Medical biochemistry, Cairo university; Mohamed M Tawfic, Study Chair — Tropical Medicine department, bny swif university; Yehia M Korriem, Study Chair — Tropical Medicine department, bny swif university; Nadia A Abdelkader, Study Chair — Tropical Medicine department, Ain Shams university; Amany Y Elkazaz, Study Chair — Medical Biochemistry, faculty of Medicine Suez Canal University; Mohamed Ghussin, Study Chair — Biochemistry department, faculty of Pharmacology Ghazza University.
Locations (2):
- Egypt (2):
  - Tropical Medicine department, Bny swif university, Bny Swif, Bny Swif
  - Medical biochemistry department, Cairo university, Cairo, Cairo Governorate